CLINICAL TRIAL: NCT03420222
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Intermittent Explosive Disorder (IED)
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Intermittent Explosive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to limited enrollment (N=10), this clinical trial was terminated by the Sponsor.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-AVP-786-206
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Intermittent Explosive Disorder
Keywords: Intermittent Explosive Disorder; AVP-786
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVP-786 (Experimental): Participants were to receive AVP-786-28 (deudextromethorphan hydrobromide [d6-DM] 28 milligrams [mg]/quinidine sulfate [Q] 4.9 mg) once daily (OD) for the first 7 days, followed by AVP-786-28 twice daily (BID) for the next 7 days. Beginning on Day 15, participants were to receive AVP-786-42.63 (d6-DM 42.63 mg/Q 4.9 mg) BID for 10 weeks.
  Interventions: Drug: AVP-786
- Placebo (Placebo Comparator): Participants were to receive placebo BID for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVP-786 — oral capsules
  Arms: AVP-786
Drug: Placebo — oral capsules
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate AVP-786 for the treatment of Intermittent Explosive Disorder (IED).

DETAILED DESCRIPTION:
Eligible participants for this study must have a diagnosis of current IED.

This is a multicenter, randomized, double-blind, placebo-controlled study, consisting of up to 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of current Intermittent Explosive Disorder (IED) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, as solicited by the Structured Clinical Interview for DSM-5, Clinical Trials Version
* At least 3 IED days (at least 1 IED episode each day, as recorded by the participant) per week for the 2 consecutive weeks directly preceding baseline with 70% compliance during that time frame, as assessed by the investigator
* Score ≥ 12 on the Life History of Aggression scale at screening
* Score ≥ 6 on the Overt Aggression Scale - Modified Total Irritability at screening and baseline
* Score ≥ 4 on the modified Clinical Global Impression of Severity for IED at screening and baseline

Exclusion Criteria:

* Diagnosis of major depressive disorder within 6 months of screening
* Significant symptoms of a depressive disorder or a Patient Health Questionnaire-9 score ≥ 10 at screening
* Met only the DSM-5 A2 criterion for IED
* Lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, antisocial personality disorder, neurocognitive disorder, or mental retardation (DSM-5 criteria)
* Recurrent IED episodes that are better explained by another mental disorder or attributable to another medical condition (e.g., head trauma, Alzheimer's disease) or to the physiological effect of a substance (e.g., a drug of abuse, a medication) (DSM-5 criteria)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Sarkis Clinical Trials, Gainesville, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - University of Chicago Medical Center Clinical Trial Site 2, Chicago, Illinois
  - BTC of New Bedford, New Bedford, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Atlea Research Institute, Las Vegas, Nevada
  - Manhattan Behavioral Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Research Institute Lindner Center of Hope/University of Cincinnati, Mason, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were screened; 27 participants were screen failures, and 10 were randomized to treatment.
Groups:
- AVP-786: Participants received AVP-786-28 (deudextromethorphan hydrobromide [d6-DM] 28 milligrams [mg]/quinidine sulfate [Q] 4.9 mg) once daily (OD) for the first 7 days, followed by AVP-786-28 twice daily (BID) for the next 7 days. Beginning on Day 15, participants received AVP-786-42.63 (d6-DM 42.63 mg/Q 4.9 mg) BID for 10 weeks.
- Placebo: Participants received placebo BID for 12 weeks.
Period: Overall Study
Arm/Group | AVP-786 | Placebo
Started | 8 | 2
Completed | 3 | 1
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AVP-786 | Placebo | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA (NA) — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA (NA) — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Baseline data have not been reported due to the low number of enrolled participants and the increased risk of patient identification. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Overt Aggression Scale - Modified for Outpatient Use (OAS-M) Total Aggression Score at Week 12
Description: The OAS-M is a clinical-administered instrument designed to assess various manifestations of aggressive behavior through 2 domains: aggression and irritability. The OAS-M aggression domain includes 4 items: verbal assault, assault against objects, assault against others, and assault against self. The rater determines the frequency of each response (item) during the past week, and the frequency of each item is multiplied by the severity level (0 to 5), producing a raw score. This raw score is multiplied by severity weight for that item (verbal assault x 1, assault against objects x 2, assault against others x 3, and assault against self x 3). Each response is scored using a 6-point scale (0 = no events to 5 = most severe form of assault within that category). The weighted individual item scores are added to obtain the OAS-M Total Aggression score. Higher scores indicate increased aggression.
Time Frame: Baseline; Week 12
Population: As the study was terminated early due to a business decision, with lack of enrollment, the data for this outcome measure was not collected or analyzed as planned.
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in the OAS-M Total Irritability Score at Week 12
Description: The OAS-M is a clinical-administered instrument designed to assess various manifestations of aggressive behavior through 2 domains: aggression, and irritability. The OAS-M irritability domain includes 2 global assessment items: global subjective irritability and global overt irritability. Each response is scored using a 6-point scale (0 = not at all to 5 = extreme). The 2 scores are added to create the OAS-M Total Irritability score (range = 0 to 10). Higher scores indicate increased irritability.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in the OAS-M Individual Items for Aggression at Week 12
Description: The OAS-M is a clinical-administered instrument designed to assess various manifestations of aggressive behavior through 2 domains: aggression and irritability. The OAS-M aggression domain includes 4 items: verbal assault, assault against objects, assault against others, and assault against self. The rater determines the frequency of each response (item) during the past week, and the frequency of each item is multiplied by the severity level (0 to 5), producing a raw score. This raw score is multiplied by severity weight for that item (verbal assault x 1, assault against objects x 2, assault against others x3, and assault against self x 3). Each response is scored using a 6-point scale (0 = no events to 5 = most severe form of assault). Higher scores indicate increased aggression.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in the OAS-M Individual Items for Irritability at Week 12
Description: The OAS-M is a clinical-administered instrument designed to assess various manifestations of aggressive behavior through 2 domains: aggression and irritability. The OAS-M irritability domain includes 2 items: global subjective irritability and global overt irritability. Each response is scored using a 6-point scale (0 = not at all; 5 = extreme). Higher scores indicate increased irritability.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in the Number of Intermittent Explosive Disorder (IED) Days Documented by Participants at Week 12
Description: The IED episodes were to be documented by the participants each evening before bedtime.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in the Number of IED Days as Assessed by the Investigator at Week 12
Description: The IED episodes were to be documented by the participants each evening before bedtime and reviewed by the Investigator post dose.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in the Number of IED Episodes at Week 12
Description: The IED episodes were to be documented by the participants each evening before bedtime. If the participant indicated that he/she experienced an IED episode, he/she was to document the number of episodes.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in the Severity of IED Episodes at Week 12
Description: The IED episodes were to be documented by the participants each evening before bedtime. If the participant indicated that he/she experienced an IED episode, he/she was to document the number of episodes and to rate the severity of the worst episode (0 = not severe at all to 10 = worst severity imaginable).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in the Severity of Distress From Episodes at Week 12
Description: The IED episodes were to be documented by the participants each evening before bedtime. If the participant indicated that he/she experienced an IED episode, he/she was to document the number of episodes and to rate the severity of distress experienced by the episode(s) (0 = no distress to 10 = worst distress imaginable).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in the OAS-M: Number of Discrete IED Episodes at Week 12
Description: The OAS-M is a clinical-administered instrument designed to assess various manifestations of aggressive behavior through 2 domains: aggression, and irritability. The OAS-M includes information regarding the number of Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) A1 aggressive episodes, and the number of DSM-5 A2 aggressive episodes experienced by the participants during the past week. The number of discrete IED episodes is calculated after an interview with the participant. Episodes identified as discrete are separated by at least 30 minutes; episodes separated by less than 30 minutes are considered a single episode.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in the Modified Clinical Global Impression of Severity (mCGI-S) Score for IED at Week 12
Description: The mCGI-S is a modified version of the CGI-S scale that provides a global evaluation of the participant's IED symptoms (e.g., aggression, anger, and irritability). The mCGI-S scale measures the severity of the participant's symptoms from the clinician's perspective in the context of other participants with IED. The mCGI-S responses are scored on a 7- point scale (1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in the Modified Clinical Global Impression of Change (mCGI-C) Score for IED at Week 12
Description: The mCGI-C is a modified version of the CGI-C scale. The clinician rates the overall global change in the participant's IED symptoms (e.g., aggression, anger, and irritability) from Baseline at the scheduled double- blind visits. The mCGI-C responses are scored using a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in the Modified Patient Global Impression of Severity (mPGI-S) Score for IED at Week 12
Description: The mPGI-S is a single-question scale. Participants rate the overall global severity of their IED symptoms (e.g., aggression, anger, and irritability) using a 7-point scale (1 = normal, no symptoms; 2 = borderline symptoms; 3 = mild symptoms; 4 = moderately bad symptoms; 5 = markedly bad symptoms; 6 = severely bad symptoms; 7 = extremely bad symptoms).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in the Modified Patient Global Impression of Change (mPGI-C) Score for IED at Week 12
Description: The mPGI-C is a single-question scale. Participants rate the overall global change in their IED symptoms (e.g., aggression, anger, and irritability) from Baseline at the scheduled double-blind visits. The mPGI- C responses are scored using a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Score at Week 12
Description: The SDS is a 3-item, participant-rated questionnaire used to evaluate impairments in the domains of work/school, social life or leisure activities, and family life or home responsibility. Participants rate the degree of impairment in work/school, social life or leisure activities, and family life or home responsibility as a result of IED symptoms using a visual analogue scale (0 = no impairment; 1, 2, 3 = mildly; 4, 5, 6 = moderately; 7, 8, 9 = markedly; 10 = extremely). Only those score categories with at least one participant with event are reported.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in the Short-Form 12-Item Health Survey (SF-12) Score at Week 12
Description: The SF-12 is a 12-item, participant self-rated questionnaire used to measure the general health status and quality of life. The SF-12 includes questions to measure the effects of health on physical functioning, role limitations due to physical health, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores range from 0 to 100. Higher scores indicate better health status.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in the State-Trait Anger Expression Inventory-2 (STAXI-2) Score at Week 12
Description: The STAXI-2 is a 57-item, participant self-rated scale used to measure the intensity of anger as an emotional state (state anger) and the disposition to experience angry feelings as a personality trait (trait anger). The STAXI-2 includes a measure of state anger, trait anger, anger expression-out, anger expression-in, anger control-out and anger control, and the anger expression index (an overall measure of the expression and control of anger). The state anger items are scored using a 4-point scale (1 = not at all to 4 = very much so) to assess the intensity of anger feelings at a particular moment. The other scales are scored using a 4- point scale to assess how frequently angry feelings are experienced, expressed, suppressed, or controlled (1 = almost never to 4 = almost always).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Arm/Group | AVP-786 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 85
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred after the first dose of the study drug through 30 days after the last dose. TEAEs are reported for all participants who received study medication. Participants were included in the treatment group based on the actual treatment received.
Arm/Group | AVP-786 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 4/8 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-786 (N=8) | Placebo (N=2)
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to limited enrollment (N=10), this clinical trial was terminated by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03420222/Prot_SAP_000.pdf